CLINICAL TRIAL: NCT01671475
Title: Impact of microEEG on Clinical Management and Outcomes of Emergency Department (ED) Patients With Altered Mental Status
Brief Title: Putting Electroencephalography (EEG) in the Emergency Department
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bio-Signal Group Corp. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); State University of New York - Downstate Medical Center (Other); Kings County Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EDEEG; RC3NS070658 (NIH)
Record Dates: First submitted 2012-08-04; First posted 2012-08-23 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Altered Mental Status
Keywords: Altered Mental Status; Non-convulsive seizure; Electroencephalography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine care plus microEEG (Experimental): Subjects allocated to this group will undergo an EEG using microEEG device in addition to their routine care. The microEEG device will be used with commercially available electrodes in a headpiece configuration.
  Interventions: Device: microEEG (Bio-Signal microEEG)
- Routine care only (control group) (No Intervention): Subjects allocated to the control group will receive routine care without microEEG. The treating physician may request a standard EEG, which will be performed by the hospital EEG laboratory, if available.

INTERVENTIONS:
Device: microEEG (Bio-Signal microEEG) — At the core, the Bio-Signal microEEG, is an FDA approved miniature, battery-operated, multi-channel, and portable system that records wideband bioelectric signals. The microEEG combines the characteristics of low noise and small size, due to a number of fundamental design characteristics. It records, amplifies, and digitizes the signals at a point very close to the electrodes. This allows the length of the wires between electrodes and the recorder's amplifiers to be very short, keeping them out of the way. Short wires also reduce any inconvenience signal artifacts or other problems that may be associated with the length of the wires. The microEEG's dimensions are about 2"x2"x1".
  Arms: Routine care plus microEEG

SUMMARY:
The proposed study aims to test the impact of microEEG on clinical management (diagnosis and treatment) of emergency department patients with Altered Mental Status (AMS). The study will utilize a portable, wireless, FDA-approved device (microEEG) as the intervention. Patients will be randomized to routine care plus microEEG (experimental arm) or routine care alone (control arm). The investigators hypothesize that incorporating microEEG in the work up of patients with AMS will impact the clinical management of these patients.

DETAILED DESCRIPTION:
Approximately, 4% and 10% of emergency department (ED) patients in the United States present with altered mental status (AMS). According to previous studies, close to 30% of AMS cases occur due to neurological etiologies. Among these pathologies are non-convulsive seizures (NCS) and non-convulsive status epilepticus (NCSE). In our previous study, the investigators established that approximately 4% (95% confidence interval, 2-8%) of ED patients with AMS suffer from NCS and NCSE. Our study also revealed that 78% of the ED patient with AMS have some form of EEG abnormality.

NCS and NCSE are difficult to diagnose especially in AMS patients because performing a thorough physical examination or obtaining medical history is often impossible in altered patients. Definitive diagnosis of NCS/NCSE requires electroencephalography (EEG), a test that records brain electrical activity and provides information about the brain function.

Unfortunately, obtaining an EEG in the ED can be challenging. This requires transporting an EEG machine to patient's bedside, where space limitations and presence of variety of monitors and devices, especially in over-crowded EDs render this practice difficult. In many institutions an EEG service is not offered after work hours due to the unavailability of 24/7 EEG technologist coverage and real-time electroencephalographer interpretation. As a result of the aforementioned limitations, ED physicians may refrain from ordering EEG.

The wireless portable EEG device (microEEG) designed by the Bio-Signal Group was designed to address these limitations. With minimal training, ED personnel could use this small, microEEG device to obtain an EEG. The recording then can be wirelessly transmitted to a host computer via a secure network connection to the neurology experts who could interpret the EEG. Incorporating microEEG in the initial workup of patients with AMS could help the ED attending rule out NCS/NCSE and focus on other diagnoses. Alternatively, if the presence of NCS is confirmed by EEG, the treatment could be initiated early and potentially reduce morbidity or mortality.

The investigators hypothesize that incorporating EEG in the work of ED patients with AMS could impact the management(diagnosis and treatment)of these patients and influence their clinical outcome.

Sample size: Our sample size analysis using data one published related study reveled that the study would need 65 patients in each group (total n:130). However, the investigators plan to perform an interim analysis after enrolling half of this target sample and adjust the sample size calculation based on the collected data if necessary.

ELIGIBILITY:
Inclusion Criteria:

ED patients ≥ 18 years old with AMS.

Exclusion Criteria:

1. Patients with apparent and immediately correctable cause of AMS (determined by ED attending during initial evaluation) that include:

   * Fingerstick or serum glucose less than 60mg/dl
   * Hypothermia (Hypothermia is defined as any body temperature below 35.0 C [95.0 F]).
   * Hyperthermia, heat exhaustion or heat stroke
   * Opioid overdose responding to Narcan.
2. Patients who cannot undergo EEG recordings for any reason (e.g. severe scalp injury).
3. Hemodynamically unstable patients(SBP <90mm Hg)
4. Patients who are uncooperative or combative.
5. Patients transferred out of ED before enrollment.
6. Patients with obvious tonic-clonic or focal seizures in the ED.

Note: Patients with hypoglycemia who do not return to their baseline level of mental status within 30 minutes of correcting their blood glucose level, will be enrolled. Similarly, patients who had an obvious seizure in the ED but do not return to their baseline mental status within 15 minutes will also be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change of ED management | 4-6 hours of arrival
  Primary outcome: Change in management (Diagnosis and Therapy)

SECONDARY OUTCOMES:
Other Outcomes | From date of randomization until the date of discharge from the hospital or date of in-hospital death from any cause, whichever comes first, assessed up to 90 days
  Secondary Outcome: Length of stay in Hospital, Length of stay in ED, In-hospital mortality, Type of ED Disposition and Type of hospital disposition.

CONTACTS AND LOCATIONS:
Overall Officials: Shahriar Zehtabchi, MD, Principal Investigator — Physician
Locations (2):
- United States (2):
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brookyln, New York

REFERENCES:
- [Derived] Zehtabchi S, Abdel Baki SG, Omurtag A, Sinert R, Chari G, Roodsari GS, Weedon J, Fenton AA, Grant AC. Effect of microEEG on clinical management and outcomes of emergency department patients with altered mental status: a randomized controlled trial. Acad Emerg Med. 2014 Mar;21(3):283-91. doi: 10.1111/acem.12324. PMID 24628753